CLINICAL TRIAL: NCT05649566
Title: Intervention of Virtual Reality on Oculomotor Muscles and Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escoles Universitaries Gimbernat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VRoculomotor
Record Dates: First submitted 2022-11-30; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Postural Balance
Keywords: Postural Balance; Oculomotor Muscles; Virtual Reality

STUDY DESIGN:
Intervention Model Description: A clinical trial is proposed with young men and women between 18 and 25 years old and physically active (targeted with the International Physical Activity Questionnaire, IPAQ).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Game Group (Experimental): A total of 24 interventions will be carried out for each participant, separated by 2 each week for 3 months. Each intervention will consist of a VR session lasting 30 minutes. Each participant must play for 30 minutes in the game "Beat know". The game consists of cutting mobile targets, using lightsabers while avoiding obstacles that approach the user. This game is a reference for immersive play since, while distracting, it recreates a physical activity similar to what would be done in reality. It has been shown that the same energy expenditure, on the part of the user, practicing tennis in real life, is what he does playing "Beat Saber" playing the same period of time.
  Interventions: Device: Virtual Reality game
- Control Group (No Intervention): No intervention during 12 weeks.

INTERVENTIONS:
Device: Virtual Reality game — The game consists of cutting mobile targets, using lightsabers while avoiding obstacles that approach the user. This game is a reference for immersive play since, while distracting, it recreates a physical activity similar to what would be done in reality. It has been shown that the same energy expenditure, on the part of the user, practicing tennis in real life, is what he does playing "Beat Saber" playing the same period of time.
  Other Names: Beat Saber on Oculus Quest 2 glasses
  Arms: Virtual Reality Game Group

SUMMARY:
Prospective, controlled, randomized, non-masked longitudinal research project for the realization of a doctoral thesis, based on an intervention with virtual reality in order to assess whether the influence on balance and the oculomotor muscles is positive.

The introduction of new technologies in the field of medicine in all fields, and in particular the rehabilitation is fully in place and under development. There are numerous examples like these technologies, including virtual reality (VR), have helped different health fields such as surgery or physiotherapy.

The main aim of the study is to analyze these factors and analyze the way in which virtual reality (VR) can modulate the convergence of the gaze and can influence the center of pressure (COP). As secondary objectives es proposes to analyze the interrelationship between the VR and the COP to analyze the clinical possibilities of application in the field of rehabilitation, whether due to a downward (oculomotor) or upward alteration (COP alteration), as well as if physical activity or gender can also influence.

DETAILED DESCRIPTION:
The center of pressure (COP) is the point where the resultant of the ground reaction forces is applied to the base of support. The oscillation of the individual with respect to the ground is projected in an anteroposterior line (AP) and another mediolateral (ML). With these two parameters you can define the total route covered by the COP. The population general presents a small area: parameters of short distance and fast and precise displacements. An alteration of the balance can be objectified by measuring an increase in the same area; reflecting a loss of axis control AP and ML and a slowing in the perception of this loss.

The oculomotor muscles are responsible for maintaining horizontal gaze; given the position bipedal, the brain seeks to maintain this premise to allow carrying out the usual activities in it position A good response of this musculature, specifically, the ability to accommodate the convergence of the look, will guarantee optimal function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 years old.
* No visual alteration.
* No history of vertigo.
* No pathology that compromises balance.
* Physically active (where the first two questions are affirmative and are 3 days and 3 hours, respectively.

Exclusion Criteria:

* Taking medication that affects the nervous and/or motor system.
* Smoking, alcoholism, taking illicit drugs or neurologically active medications.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Centre Of Pressure at 7 days after 12th session | Day 1 and 7 days after the 12th session.
  The pressure center (COP) is the point where the resulting reaction forces with the ground is applied to the support base. The oscillation of the individual with respect to the ground is projected in an anteroposterior line (AP) and a mediolateral line (ML). With these two parameters, the total route covered by the COP can be defined. An alteration of balance can be objectified by measuring an increase in the same area; reflecting a loss of control of the AP and ML axes and a slowdown in the perception of this loss.

SECONDARY OUTCOMES:
Change from Baseline PPC at 7 days after 12th session | Day 1 and 7 days after the 12th session.
  The Near Convergence Point (PPC) test analyzes the effectiveness of the oculomotor muscles, consists of showing a stimulus 40 centimeters from the participant, a point where the vision of this stimulus should not be double. The stimulus will approach until the participant sees double, it is the breaking point and it will be the PPC to be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Gomez Doctor, PT, MsC, Principal Investigator — E.U. Gimbernat
Locations (1):
- Escoles Universitaries Gimbernat, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winter, D.A., Human balance and posture control during standing and walking. Gait & Posture, 1995. 3(4): 193-214.
- [Background] León-Molina, P., et al., Center of plantar pressure and postural balance depending on the skull preposition. Rev Fac Odontol Univ Antioq 2016. 28(1): 112-122.
- [Background] Alexander NB, Galecki AT, Nyquist LV, Hofmeyer MR, Grunawalt JC, Grenier ML, Medell JL. Chair and bed rise performance in ADL-impaired congregate housing residents. J Am Geriatr Soc. 2000 May;48(5):526-33. doi: 10.1111/j.1532-5415.2000.tb04999.x. PMID 10811546
- [Background] Cheng PT, Wu SH, Liaw MY, Wong AM, Tang FT. Symmetrical body-weight distribution training in stroke patients and its effect on fall prevention. Arch Phys Med Rehabil. 2001 Dec;82(12):1650-4. doi: 10.1053/apmr.2001.26256. PMID 11733877
- [Background] Brandt T, Krafczyk S, Malsbenden I. Postural imbalance with head extension: improvement by training as a model for ataxia therapy. Ann N Y Acad Sci. 1981;374:636-49. doi: 10.1111/j.1749-6632.1981.tb30907.x. PMID 6978651
- [Background] Jackson RT, Epstein CM. Effect of head extension on equilibrium in normal subjects. Ann Otol Rhinol Laryngol. 1991 Jan;100(1):63-7. doi: 10.1177/000348949110000110. PMID 1985528
- [Background] Paulus WM, Straube A, Brandt T. Visual stabilization of posture. Physiological stimulus characteristics and clinical aspects. Brain. 1984 Dec;107 ( Pt 4):1143-63. doi: 10.1093/brain/107.4.1143. PMID 6509312
- [Background] Pinsault N, Vuillerme N. Differential postural effects of plantar-flexor muscle fatigue under normal, altered and improved vestibular and neck somatosensory conditions. Exp Brain Res. 2008 Oct;191(1):99-107. doi: 10.1007/s00221-008-1500-z. Epub 2008 Jul 29. PMID 18663436
- [Background] Blanchet M, Prince F, Messier J. Development of postural stability limits: Anteroposterior and mediolateral postural adjustment mechanisms do not follow the same maturation process. Hum Mov Sci. 2019 Feb;63:164-171. doi: 10.1016/j.humov.2018.11.016. Epub 2018 Dec 14. PMID 30557794
- [Background] Whitney SL, Roche JL, Marchetti GF, Lin CC, Steed DP, Furman GR, Musolino MC, Redfern MS. A comparison of accelerometry and center of pressure measures during computerized dynamic posturography: a measure of balance. Gait Posture. 2011 Apr;33(4):594-9. doi: 10.1016/j.gaitpost.2011.01.015. Epub 2011 Feb 17. PMID 21333541
- [Background] Winter, David A. Review Article: Human balance and posture control during standing and walking. Gait and posture, 1995. 3: p 193-214
- [Background] Chandler JM, Duncan PW, Studenski SA. Balance performance on the postural stress test: comparison of young adults, healthy elderly, and fallers. Phys Ther. 1990 Jul;70(7):410-5. doi: 10.1093/ptj/70.7.410. PMID 2192373
- [Background] Sofianidis G, Dimitriou AM, Hatzitaki V. A Comparative Study of the Effects of Pilates and Latin Dance on Static and Dynamic Balance in Older Adults. J Aging Phys Act. 2017 Jul;25(3):412-419. doi: 10.1123/japa.2016-0164. Epub 2017 Jun 28. PMID 27992251
- [Background] Mestre C, Bedell HE, Diaz-Douton F, Pujol J, Gautier J. Characteristics of saccades during the near point of convergence test. Vision Res. 2021 Oct;187:27-40. doi: 10.1016/j.visres.2021.06.001. Epub 2021 Jun 17. PMID 34147850
- [Background] Erhardsson M, Alt Murphy M, Sunnerhagen KS. Commercial head-mounted display virtual reality for upper extremity rehabilitation in chronic stroke: a single-case design study. J Neuroeng Rehabil. 2020 Nov 23;17(1):154. doi: 10.1186/s12984-020-00788-x. PMID 33228710
- [Background] Rutkowski S, Adamczyk M, Pastula A, Gos E, Luque-Moreno C, Rutkowska A. Training Using a Commercial Immersive Virtual Reality System on Hand-Eye Coordination and Reaction Time in Young Musicians: A Pilot Study. Int J Environ Res Public Health. 2021 Feb 1;18(3):1297. doi: 10.3390/ijerph18031297. PMID 33535539
- [Background] Prasertsakul T, Kaimuk P, Chinjenpradit W, Limroongreungrat W, Charoensuk W. The effect of virtual reality-based balance training on motor learning and postural control in healthy adults: a randomized preliminary study. Biomed Eng Online. 2018 Sep 18;17(1):124. doi: 10.1186/s12938-018-0550-0. PMID 30227884
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Minoonejad H, Barati AH, Naderifar H, Heidari B, Kazemi AS, Lashay A. Effect of four weeks of ocular-motor exercises on dynamic visual acuity and stability limit of female basketball players. Gait Posture. 2019 Sep;73:286-290. doi: 10.1016/j.gaitpost.2019.06.022. Epub 2019 Jul 16. PMID 31398634
- [Background] Szpak A, Michalski SC, Loetscher T. Exergaming With Beat Saber: An Investigation of Virtual Reality Aftereffects. J Med Internet Res. 2020 Oct 23;22(10):e19840. doi: 10.2196/19840. PMID 33095182
- [Background] Alsiri N, Cramp M, Barnett S, Palmer S. Gait biomechanics in joint hypermobility syndrome: a spatiotemporal, kinematic and kinetic analysis. Musculoskeletal Care. 2020 Sep;18(3):301-314. doi: 10.1002/msc.1461. Epub 2020 Feb 22. PMID 32086882
- [Background] Lai B, Davis D, Narasaki-Jara M, Hopson B, Powell D, Gowey M, Rocque BG, Rimmer JH. Feasibility of a Commercially Available Virtual Reality System to Achieve Exercise Guidelines in Youth With Spina Bifida: Mixed Methods Case Study. JMIR Serious Games. 2020 Sep 3;8(3):e20667. doi: 10.2196/20667. PMID 32880577
- [Background] Ernst N, Schatz P, Trbovich AM, Emami K, Eagle SR, Mucha A, Collins MW, Kontos AP. Utility of 1 Measurement Versus Multiple Measurements of Near Point of Convergence After Concussion. J Athl Train. 2020 Aug 1;55(8):850-855. doi: 10.4085/1062-6050-431-19. PMID 32577736